CLINICAL TRIAL: NCT02924766
Title: A Safety and Pharmacokinetics Study of Niraparib Plus Androgen Receptor-Targeted Therapy (Apalutamide or Abiraterone Acetate Plus Prednisone) in Men With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Safety and Pharmacokinetics Study of Niraparib Plus an Androgen Receptor-Targeted Therapy in Men With Metastatic Castration-Resistant Prostate Cancer (BEDIVERE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108230; 2016-002694-35 (EudraCT Number); 64091742PCR1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — niraparib; apalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Niraparib + Apalutamide/[Abiraterone Acetate + Prednisone] (Experimental): Participants will receive initial starting dose of Niraparib 200 milligram (mg) once daily in combination either with Apalutamide 240 mg (4*60 mg) once daily or Abiraterone Acetate 1000 mg (4*250 mg) plus 10 mg Prednisone (5 mg twice daily) for 28 days of cycle 1. Once a safe dose of niraparib is selected with each Andrgen Receptor (AR)-targeted therapy [Apalutamide or Abiraterone Acetate plus Prednisone], then an expansion phase (Part 2) will open to further explore safety and assess antitumor activity.
  Interventions: Drug: Niraparib; Drug: Apalutamide; Drug: Abiraterone Acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Niraparib — Participants will start with niraparib 200 mg once daily.
  Other Names: JNJ-64091742
Drug: Apalutamide — Participants will receive apalutamide 240 mg (4*60 mg) once daily orally.
  Other Names: ARN-509
Drug: Abiraterone Acetate — Participants will receive 1000 mg (4*250mg) once daily.
  Other Names: ZYTIGA
Drug: Prednisone — Participants will receive 10 mg (1*5 mg twice daily).

SUMMARY:
The purpose of this study is to assess the safety and pharmacokinetics of niraparib when administered in combination with an androgen receptor (AR)-targeted therapy (apalutamide or abiraterone acetate plus prednisone) in adult men with metastatic castration resistant prostate cancer (mCRPC) who may or may not have deoxyribonucleic acid (DNA)-repair anomalies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer (mixed histology is acceptable, with the exception of the small cell pure phenotype, which is be excluded
* At least 1 line of prior taxane-based chemotherapy
* At least 1 line of prior androgen receptor (AR) targeted therapy
* Progression of metastatic prostate cancer in the setting of castrate levels of testosterone or history of bilateral orchiectomy at study entry
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of lesser than or equal to [<=]1

Exclusion Criteria:

* Known brain metastases or history of seizure
* Prior treatment with a poly (adenosine diphosphate [ADP] ribose) polymerase (PARP) inhibitor
* Prior platinum-based chemotherapy for the treatment of prostate cancer
* Known history or current diagnosis of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Severe or unstable cardiovascular disease or uncontrolled hypertension
* Left ventricular ejection fraction (LVEF) of lesser than [<] 50 percent (%) as determined by multiple uptake gated acquisition (MUGA) or echocardiography during screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Determine Recommended Phase 2 dose (RP2D) of Niraparib in Combination With 240 milligram (mg) Apalutamide or 1,000 mg Abiraterone Acetate Plus 10 mg Prednisone (5 mg Twice Daily) in Part 1 | Up to 56 days
  RP2D will be defined as the highest dose of study drug at which less than 33 percent (%) of participants experience dose limiting toxicity (DLT).
Number of Participants With Incidence and Severity of Adverse Events (Part 2) | Up to 30 days after last dose
  Number of participants will be assessed to further explore safety and antitumor activity in Part 2 (dose expansion) of study.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 24 hours postdose on Cycle 1 Day 1 up to 10 hours postdose Cycle 3 Day 1 (each cycle 28 days)
  Maximum observed plasma concentration (Cmax) will be assessed.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) | 24 hours postdose on Cycle 1 Day 1 up to 10 hours postdose Cycle 3 Day 1 (each cycle 28 days)
  Time to reach the maximum plasma concentration(Tmax) will be assessed.
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC [0-24]) | 24 hours postdose on Cycle 1 Day 1 up to 10 hours postdose Cycle 3 Day 1 (each cycle 28 days)
  Area under plasma concentration-time curve from time 0 to time 24 hours after dosing will be assessed.
Trough Plasma Concentration (Ctrough) | Predose (Cycle 1 Days 15 and 22) up to Cycle 3 Day 1 (each cycle 28 days) then Every 3 Cycles after Cycle 3 till End of Treatment (30 days after last dose)
  Ctrough is the minimum observed (that is, predose) plasma concentration following multiple dosing will be assessed.
Metabolite to Parent Ratio for Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC [0-24]) | 24 hours postdose on Cycle 1 Day 1 up to 10 hours postdose Cycle 3 Day 1 (each cycle 28 days)
  Metabolite to parent drug ratio for area under the plasma concentration-time curve from time 0 to 24 hours (AUC [0-24]) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- United States (4):
  - West Hollywood, California
  - Louisville, Kentucky
  - Portland, Oregon
  - Myrtle Beach, South Carolina
- Canada (2):
  - Vancouver, British Columbia
  - Montreal, Quebec

REFERENCES:
- [Derived] Saad F, Chi KN, Shore ND, Graff JN, Posadas EM, Lattouf JB, Espina BM, Zhu E, Yu A, Hazra A, De Meulder M, Mamidi RNVS, Bradic B, Francis P, Hayreh V, Rezazadeh Kalebasty A. Niraparib with androgen receptor-axis-targeted therapy in patients with metastatic castration-resistant prostate cancer: safety and pharmacokinetic results from a phase 1b study (BEDIVERE). Cancer Chemother Pharmacol. 2021 Jul;88(1):25-37. doi: 10.1007/s00280-021-04249-7. Epub 2021 Mar 22. PMID 33754187
- See also: A Safety and Pharmacokinetics Study of Niraparib plus Androgen Receptor-Targeted Therapy (Apalutamide or Abiraterone Acetate plus Prednisone) in Men with Metastatic Castration-Resistant — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108230&attachmentIdentifier=6859793c-4a76-466e-ad41-843b583b6c9c&fileName=CR108230_CSR_Synopsis.pdf&versionIdentifier=